CLINICAL TRIAL: NCT04441671
Title: Oral Disodiumpyrophosphate (Na2H2PPi) Absorption in Pseudoxanthoma Elasticum (PXE)
Brief Title: Oral Pyrophosphate Absorption in PXE Disease
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Withdrawn
Sponsor: Tampere University Hospital (Other)
Collaborators: UMC Utrecht (Other); Hungarian Academy of Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R19017M; 2019-002109-24 (EudraCT Number); KLnro 38/2019 (Other: Fimea)
Record Dates: First submitted 2020-01-20; First posted 2020-06-22 (Actual); Last update posted 2021-04-22 (Actual); Status verified 2021-04

CONDITIONS: Pseudoxanthoma Elasticum
MeSH Terms: conditions — Pseudoxanthoma Elasticum | interventions — sodium pyrophosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Open label (Experimental): Disodiumpyrophosphate, capsuled powder, First day: 30 mg/kg fasting at 08.00 and with standard mixed meal at 12.00 Second day: 50 mg/kg fasting at 08.00 and with standard mixed meal at 12.00
  Interventions: Drug: Disodium Pyrophosphate

INTERVENTIONS:
Drug: Disodium Pyrophosphate — Absorption trial
  Other Names: Na2H2PPi

SUMMARY:
Pyrophosphate is an endogenous, non-toxic metabolite inhibiting soft tissue calcification. The aim of our study is to find optimal dosing and safety of oral disodium-PPi (Na2H2PPi). Absorption curves (pharmacokinetics), AUC0-t, Cmax and Tmax for PPi and phosphate will be provided for healthy controls and PXE-patients both fasting and with standard meal intake.

DETAILED DESCRIPTION:
Phase II oral capsulized disodium-PPi (Na2H2PPi) powder absorption study in subjects with PXE (n=8-12) will be done in the ward of Internal Medicine of Tampere University Hospital and University Medical Center Utrecht.

After a 10-hour fast at 8.00 a.m. 30 mg/kg (first day) and 50 mg/kg (second day) capsulized dose of PPi will be given with 2 dl water. At 12.00 a.m. another capsulized 30 mg/kg (first day) or 50 mg/kg (second day) single dose of PPi with a standard mixed meal (lunch) will be given with 2 dl water at the time when a subject starts eating.

Plasma and urine sampling include plasma and spot urine electrolytes, creatinine, and pyrophosphate. Plasma sampling will be done at 0, 15, 30, 60, 120 and 240 min after ingestion of PPi. Urine spot sample will be taken at 0 and 240 min after ingestion of PPi.

Physical activity is restricted. Side-effects will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Adults (>18 yrs)
* clinically and genetically proven PXE
* Body mass index (BMI) 18,5-34,9 kg/m2

Exclusion Criteria:

* Special groups according to researchers' decision.
* Pregnancy
* No effective contraception in females in child-bearing age.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-12-08 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Concentration area under the curve 0-t of pyrophosphate | two days
Maximal concentration of pyrophosphate | two days
  Cmax
Timepoint of maximal pyrophosphate concentration | two days
  Tmax

SECONDARY OUTCOMES:
Concentration area under the curve 0-t of phosphate | two days
  AUC0-t
Maximal concentration of phosphate | two days
  Cmax
Timepoint of maximal phosphate concentration | two days
  Tmax

CONTACTS AND LOCATIONS:
Overall Officials: Pasi I Nevalainen, MD, PhD, Principal Investigator — Tampere University Hospital

IPD SHARING:
Plan to Share IPD: No
Only anonymized data can be shared